CLINICAL TRIAL: NCT01640314
Title: A Phase 3 Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, Influenza Vaccine Produced in Mammalian Cell Culture (Optaflu®), Formulation 2012/2013, When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of a Cell Derived Subunit Trivalent Nonadjuvated Influenza Study Vaccine in Adults Aged 18 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V58_32S; 2011-006277-25 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-07-13 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
Keywords: Influenza; Adults; Elderly; Immunology; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cell derived subunit trivalent nonadjuvanted vaccine (Experimental)
  Interventions: Biological: Cell derived subunit trivalent nonadjuvanted vaccine

INTERVENTIONS:
Biological: Cell derived subunit trivalent nonadjuvanted vaccine — A single 0.5 mL dose of the cell derived subunit trivalent nonadjuvated influenza vaccine (TIVc) supplied in prefilled syringes and administered intramuscularly in the deltoid muscle (preferably) of the non dominant arm.

SUMMARY:
The purpose of this study is to evaluate the safety of a single intramuscular (IM) injection of the cell derived subunit trivalent nonadjuvanted influenza vaccine in adult and elderly subjects and the antibody response to each influenza vaccine antigen, as measured by hemagglutination inhibition (HI) at approximately 21 days postimmunization in adult and elderly subjects in compliance with the requirements of the current EU recommendations for clinical trials related to yearly licensing of influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers of 18 years of age or older;
2. Individuals able to comply with all the study requirements;
3. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
2. Individuals with any serious chronic or acute disease (in the judgment of the investigator), including but not limited to:

   * Medically significant cancer (except for benign or localized skin cancer, cancer in remission for ≥10 years or localized prostate cancer that has been clinically stable for more than 2 years without treatment);
   * Medically significant advanced congestive heart failure (ie. NYHA class III and IV);
   * Chronic obstructive pulmonary disease (COPD; i.e., GOLD Stage III and IV);
   * Autoimmune disease (including rheumatoid arthritis, except for Hashimoto's thyroiditis that has been clinically stable for ≥5 years);
   * Diabetes mellitus type I;
   * Poorly controlled diabetes mellitus type II;
   * Advanced arteriosclerotic disease;
   * History of underlying medical condition such as major congenital abnormalities requiring surgery, chronic treatment, or associated with developmental delay (e.g., Down's syndrome);
   * Acute or progressive hepatic disease;
   * Acute or progressive renal disease;
   * Severe neurological (es. Guillain-Barré syndrome) or psychiatric disorder;
   * Severe asthma.
3. Individuals with history of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g.Influenza viral protein).
4. Individuals with known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting, for example, from:

   * receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study;
   * receipt of immunostimulants;
   * receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivatives within the past 3 months and for the full length of the study;
   * suspected or known HIV infection or HIV-related disease.
5. Individuals with known or suspected history of drug or alcohol abuse.
6. Individuals with a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject.
7. Individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study.
8. Individuals with history or any illness that, in the opinion of the investigator, pose additional risk to the subjects due to participation in the study.
9. Individuals who within the past 6 months have:

   * had any laboratory confirmed seasonal or pandemic influenza disease;
   * received any seasonal or pandemic influenza vaccine.
10. Individuals who received any other vaccine within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine during the study.
11. Individuals with any acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days.
12. Individuals that have experienced fever (i.e., axillary temperature ≥38°C) within the last 3 days of intended study vaccination.
13. Individuals participating in any clinical trial with another investigational product 4 weeks prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
14. Individuals who are part of study personnel or close family members conducting this study.
15. BMI >35 kg/m2.
16. Females who are pregnant (confirmed by positive urine pregnancy test) or nursing (breastfeeding). Females of childbearing potential who refuse to use an acceptable method of birth control for the whole duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (1):
- Bernhard Nocht Institute, Bernhard-Nocht-Strasse 74, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at one study centre in Germany.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- 18-60 Y: Subjects ≥18 years to ≤60 years of age who received one TIVc vaccination
- ≥ 61 Y: Subjects ≥61 years of age who received one TIVc vaccination
Period: Overall Study
Arm/Group | 18-60 Y | ≥ 61 Y
Started | 63 | 63
Completed | 63 | 62
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18-60 Y | ≥ 61 Y | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (11.4) | 68.0 (4.7) | 52.7 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Seroconversion or Significant Increase in HI Titer Against Each of Three Vaccine Strains After One Vaccination of TIVc
Description: Immunogenicity was measured as the percentage of subjects who achieved seroconversion or significant increase in hemagglutination inhibition (HI) titer, against each of three vaccine strains, three weeks after vaccination (day 22), evaluated using HI cell-derived antigen assay.
  As per the European (CHMP) criteria, seroconversion or significant increase in titer is defined as the percentage of subjects with a prevaccination HI titer <10 to a postvaccination HI titer ≥40; or in subjects with a prevaccination HI titer ≥10, a ≥4-fold increase in postvaccination HI antibody titer. This criterion is met according to CHMP guideline if percentage of subjects achieving seroconversion or significant increase in HI titer is >40% (≥18 years to ≤60 years) or 30% (≥61 years).
Time Frame: Day 22
Population: Analysis was done on the per-protocol (PP) set, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | 18-60 Y | ≥ 61 Y
Number analyzed (Participants) | 63 | 62
Percentages
  A/H1N1 | 73 [60 to 83] | 58 [45 to 70]
  A/H3N2 | 67 [54 to 78] | 45 [32 to 58]
  B | 63 [50 to 75] | 42 [30 to 55]

2. Primary Outcome: Geometric Mean Ratio of Subjects Against Each of Three Vaccine Strains After One Vaccination of TIVc
Description: Geometric mean ratio (GMR) of subjects was calculated as the ratio of postvaccination to prevaccination HI geometric mean titers (GMTs), directed against each of three vaccine strains, three weeks after vaccination (day 22).
  The CHMP criterion was met if the geometric mean increase (GMR, day 22/day 1) in HI antibody titer is >2.5 (≥18 years to ≤60 years) or >2.0 (≥61 years).
Time Frame: Day 22
Population: Analysis was done on the PP set.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | 18-60 Y | ≥ 61 Y
Number analyzed (Participants) | 63 | 62
Ratio
  A/H1N1 | 13 [8.75 to 20] | 5.79 [4.12 to 8.12]
  A/H3N2 | 6.38 [4.5 to 9.06] | 4.21 [2.96 to 5.97]
  B | 5.63 [4.11 to 7.7] | 3.54 [2.65 to 4.72]

3. Primary Outcome: Percentages of Subjects Who Achieved HI Titer ≥40 Against Each of Three Vaccine Strains After One Vaccination of TIVc
Description: Immunogenicity was measured as the percentage of subjects achieving HI titer ≥40 against each of three vaccine strains at baseline (day 1) and three weeks after TIVc vaccination (day 22).
  This criterion was met according to CHMP guideline if percentage of subjects achieving HI titer ≥40 is >70% (≥18 years to ≤60) or 60% (≥61 years).
Time Frame: Day 1 and 22
Population: Analysis was done on the PP set.
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | 18-60 Y | ≥ 61 Y
Number analyzed (Participants) | 63 | 62
Percentages
  A/H1N1 (Day 1) | 56 [42 to 68] | 61 [48 to 73]
  A/H1N1 (Day 22) | 98 [91 to 100] | 100 [94 to 100]
  A/H3N2 (Day 1) | 86 [75 to 93] | 85 [74 to 93]
  A/H3N2 (Day 22) | 100 [94 to 100] | 100 [94 to 100]
  B (Day 1) | 54 [41 to 67] | 40 [28 to 54]
  B (Day 22) | 98 [91 to 100] | 85 [74 to 93]

4. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Reactions (Day 1 - Day 4 Postvaccination)
Description: Safety was assessed as the number of subjects who reported solicited local and systemic reactions from day 1 up to and including day 4 after TIVc vaccination.
Time Frame: From day 1 through day 4 postvaccination
Population: Analysis was done on the safety dataset i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | 18-60 Y | ≥ 61 Y
Number analyzed (Participants) | 63 | 63
Number of subjects
  Injection site ecchymosis | 1 | 4
  Injection site erythema | 1 | 0
  Injection site swelling | 1 | 2
  Injection site induration | 0 | 2
  Injection site pain | 29 | 17
  Chills/shivering | 1 | 1
  Malaise | 5 | 2
  Myalgia | 27 | 12
  Arthralgia | 2 | 0
  Headache | 13 | 4
  Sweating | 10 | 7
  Fatigue | 15 | 7
  Fever (≥38°C) | 0 | 0

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving One Dose of TIVc.
Description: The number of subjects in both age groups reporting any unsolicited AEs between Day 1 to Day 22 after receiving one dose of TIVc.
Time Frame: Day 1 to Day 22
Population: Analysis was done on the safety set population.
Measure: Number; unit: Number of Subjects
Arm/Group | 18-60 Y | ≥ 61 Y
Number analyzed (Participants) | 63 | 63
Number of Subjects
  Any AEs | 9 | 12
  At least possibly related AEs | 5 | 7
  Serious AEs | 0 | 0
  At least possibly related SAEs | 0 | 0
  AEs leading to withdrawal | 0 | 0

ADVERSE EVENTS:
Time Frame: From day 1 through day 22
Description: Serious adverse events (SAEs) were collected from day 1 through day 22.
Arm/Group | 18-60 Y | ≥ 61 Y
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 45/63 | 30/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18-60 Y (N=63) | ≥ 61 Y (N=63)
Fatigue (General disorders) | 15 (15) | 7 (7)
Injection site haemorrhage (General disorders) | 1 (1) | 4 (4)
Injection site pain (General disorders) | 29 (29) | 17 (17)
Malaise (General disorders) | 5 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (27) | 12 (12)
Headache (Nervous system disorders) | 13 (13) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 (10) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No